CLINICAL TRIAL: NCT02706080
Title: Registry of Patient With Antithrombotic Agents Admitted to an Emergency
Brief Title: Registry of Patient With Antithrombotic Agents Admitted to an Emergency Department
Acronym: RATED Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0257
Record Dates: First submitted 2016-02-09; First posted 2016-03-11 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Antithrombotic Agents
Keywords: Antithrombotic agents; VKA; Direct Oral Anticoagulant; Antiplatelet; Bleeding; Emergency
MeSH Terms: conditions — Hemorrhage; Emergencies | interventions — Emergency Service, Hospital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Antithrombotic agents: We propose to realize a single-center prospective registry of patient under Antithrombotic agent who came to the emergency unit for any reason.
  Interventions: Other: emergency

INTERVENTIONS:
Other: emergency

SUMMARY:
Antithrombotics with antiplatelet agents, vitamin K antagonist (VKA), heparin and related substances, and new oral anticoagulants are prescribed for arterial diseases, especially in secondary prevention of embolic disease in carrier patients of heart valves and in patients with fibrillation atrial, and venous diseases, in prevention and treatment.

The prescription of these treatments is increasing especially in older patients associated with many comorbidities. Today, an estimated number of 900 000 patients under anti-vitamin K in France, and more than 1.5 million for patients on antiplatelet agents.

Venous thromboembolism (VTE) is common in the general population with an annual incidence of 10-18 cases per 10 000. The most severe form of VTE is represented by pulmonary embolism with a third of cases. Even if a large literature allows for high grade recommendations on many areas, there is still some gray areas regarding the long-term outcomes, the early evolution and tolerance of treatment, including long-term recurrence, the incidence of embolic sequelae with post-embolic pulmonary hypertension and association with other cardiovascular arterial accident (acute Coronary Syndrome, Stroke, arterial disease of the Lower Extremities ...).

The major risk of these antithrombotic is bleeding both in terms of morbidity mortality. Despite this risk, little study focuses on the exact epidemiology of bleeding associated with the use of antithrombotic. If the frequency of hemorrhagic stroke is low, some populations particularly at risk of bleeding represent the majority of serious bleeding events under VKA or anti-platelet. However, the VKA and antiplatelet agents are the first providers of hemorrhagic serious side effects drugs when looking at all national and international studies on the iatrogenic with in topped gastrointestinal bleeding and intracerebral hemorrhage (mortality of about 10 to 15%).

Moreover the recent arrival of new oral anticoagulants (Apixaban rivaroxaban, dabigatran ...) should profoundly change the management of venous thromboembolism and cardioembolic event. Because of their risk-benefit, simplicity and convenience of their prescription, the number of patients treated with these new anticoagulants were to rise rapidly. In addition, many patients deemed too "fragile" to be treated with VKA, should be treated with these treatments. These new anti-Xa and anti-IIa anticoagulants already marketed or about to be. They have the advantage over VKA: an oral way, their pharmacokinetic characteristics, absence of biological monitoring, chemical synthesis .... If it is not possible today to give the advantage to one or the other of these molecules, the choice will be directed by their pharmacokinetic characteristics, their half life, their method of disposal but also by patients co-morbidities. Although biological tests are currently available for the monitoring of these products, therapeutic solutions for severe bleeding does not exist: there is indeed no antidote for now, though the issue is finding a balance between increased therapeutic benefit and bleeding risk optimization. But hemorrhagic stroke is the most serious complications of oral anticoagulant therapy, with substantial documentation for these events occurring under VKA but little data on those occurring with the new oral anticoagulants (Apixaban rivaroxaban, dabigatran ...).

DETAILED DESCRIPTION:
We propose to realize a single-center prospective registry of patient under Antithrombotic agent who came to the emergency unit for any reason.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patient under antithrombotic agent who came in the emergency unit for any reason

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Antithrombotic agents
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
look for risk factors of bleeding events | at day 1
  The bleeding events was noted when the patient arrive in the emergency unit. For the major bleeding event, it was bleeding that was fatal or overt bleeding with a drop in haemoglobin level of at least 20 g/L or requiring transfusion of at least 2 units packed blood cells, or haemorrhage into a critical anatomical site (intracranial, gastrointestinal)
look for risk factors of major bleeding events | at day 1
  The bleeding events was noted when the patient arrive in the emergency unit. For the major bleeding event, it was bleeding that was fatal or overt bleeding with a drop in haemoglobin level of at least 20 g/L or requiring transfusion of at least 2 units packed blood cells, or haemorrhage into a critical anatomical site (intracranial, gastrointestinal)

SECONDARY OUTCOMES:
Number of death | at day 1
  - The number of death (with all cause of mortality) during the hospitalisation of the patient regarding the discharge letter of the patient
Adjudicated symptomatic recurrence of thromboembolic events | at day 1
number of symptomatic thromboembolic events | at day 1
  - the number of symptomatic thromboembolic events during the hospitalisation of the patient regarding the discharge letter of the patient
number of cardiovascular events | at day 1
  - the number of cardiovascular events during the hospitalisation of the patient regarding the discharge letter of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moustafa F, Malhomme R, Pereira B, Barres A, Saint-Denis J, Dutheil F, Batisse M, Schmidt J. Assessment of the Impact of L-Thyroxine Therapy on Bleeding Risk in Patients Receiving Vitamin K Antagonists. Clin Drug Investig. 2017 Oct;37(10):929-936. doi: 10.1007/s40261-017-0545-9. PMID 28612237